CLINICAL TRIAL: NCT02988817
Title: First-in-human, Open-label, Dose-escalation Trial With Expansion Cohorts to Evaluate Safety of Axl-specific Antibody-drug Conjugate (Enapotamab Vedotin, HuMax®-AXL-ADC) in Patients With Solid Tumors
Brief Title: Enapotamab Vedotin (HuMax-AXL-ADC) Safety Study in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCT1021-01; 2016-002243-42 (EudraCT Number); 211258 (Other: IRAS ID; UK Research Summaries Database)
Record Dates: First submitted 2016-12-01; First posted 2016-12-09 (Estimated); Results first posted 2023-01-05 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Ovarian Cancer; Cervical Cancer; Endometrial Cancer; Non Small Cell Lung Cancer (NSCLC); Thyroid Cancer; Melanoma; Sarcoma; Solid Tumors
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Carcinoma, Non-Small-Cell Lung; Thyroid Neoplasms; Melanoma; Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Enapotamab vedotin (HuMax-AXL-ADC) (Experimental): Participants in all cohorts of the trial (both in escalation and expansion phase) will be administered enapotamab vedotin (HuMax-AXL-ADC) intravenously (IV).
  Interventions: Biological: Enapotamab vedotin (HuMax-AXL-ADC)

INTERVENTIONS:
Biological: Enapotamab vedotin (HuMax-AXL-ADC) — Enapotamab vedotin (HuMax-AXL-ADC) will be administered intravenously.

SUMMARY:
The purpose of the trial is to determine the maximum tolerated dose and to establish the safety profile of HuMax-AXL-ADC in a mixed population of patients with specified solid tumors

DETAILED DESCRIPTION:
The trial consists of two parts; a dose escalation part (phase I, first in-human (FIH)) and an expansion part (phase IIa).

The dose escalation part has 2 dosing schedules: 1 dose every 3 weeks (1Q3W) dose regimen, and 3 doses every 4 weeks (3Q4W) dosing regimen.

The Expansion part of the trial will further explore the recommended phase 2 dose and dosing regimens of HuMax-AXL-ADC as determined in dose escalation part.

ELIGIBILITY:
Inclusion Criteria:

1. For the dose escalation part: Patients with selected, relapsed or refractory solid tumors who have failed available standard therapy or who are not candidates for standard therapy. For the expansion part: Patients with advanced and/or metastatic solid tumors who are not candidates for standard therapy
2. Patients must have measurable disease according to Response Evaluation Criteria In Solid Tumors (RECIST).
3. For the expansion patients must provide a tumor tissue sample from archival tissue or fresh biopsy at enrolment
4. Age ≥ 18 years.
5. Acceptable renal function
6. Acceptable liver function
7. Acceptable hematological status
8. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
9. Life expectancy of at least three months.
10. Patients, both females and males, of childbearing/reproductive potential must agree to use adequate contraception while included in the trial and for six months after the last infusion of HuMax-AXL-ADC
11. Patients must provide a signed informed consent form before any trial relates activities are carried out.

Exclusion Criteria:

1. Acute deep vein thrombosis or clinically relevant pulmonary embolism, not stable for at least 4 weeks prior to first IMP administration.
2. Have clinically significant cardiac disease
3. Known congestive heart failure and/ or a known decreased cardiac ejection fraction of < 45%. A baseline QT interval as corrected by Fridericia's formula (QTcF) > 480 msec, a complete left bundle branch block (defined as a QRS interval ≥ 120 msec in left bundle branch block form) or an incomplete left bundle branch block.
4. Uncontrolled hypertension
5. Have received granulocyte colony stimulating factor (G-CSF) or granulocyte/macrophage colony stimulating factor support 3 weeks prior to first IMP administration.
6. Have received a cumulative dose of corticosteroid > 150 mg prednisone (or equivalent doses of corticosteroids) within two weeks before the first Investigational Medicinal Product (IMP) administration.
7. History of ≥ grade 3 allergic reactions to monoclonal antibody therapy as well as known or suspected allergy or intolerance to any agent given in the course of this trial.
8. Major surgery within four weeks before first IMP administration.
9. Any history of intracerebral arteriovenous malformation, cerebral aneurysm, brain metastases or stroke.
10. Any anticancer therapy including; small molecules, immunotherapy, chemotherapy monoclonal antibodies or any other experimental drug within five half-lives but maximum four weeks before first infusion. Accepted exceptions are bisphosphonates, denosumab and gonadotropin-releasing hormone agonist or antagonist.
11. Prior therapy with a conjugated or unconjugated auristatin derivative/vinca-binding site targeting payload.
12. Radiotherapy within 14 days prior to first IMP administration.
13. Known past or current malignancy other than inclusion diagnosis, except for:

    * Cervical carcinoma of Stage 1B or less.
    * Non-invasive basal cell or squamous cell skin carcinoma.
    * Non-invasive, superficial bladder cancer.
    * Prostate cancer with a current prostate specific antigen (PSA) level < 0.1 ng/mL.
    * Breast cancer in BRCA1 or BRCA2 positive ovarian cancer patients.
    * Any curable cancer with a complete response (CR) of > 2 years duration.
14. Melanoma patients with an lactate dehydrogenase (LDH) ≥ 3 x upper limit normal (ULN).
15. Ongoing significant, uncontrolled medical condition including:

    o Serious, non-healing wound, skin ulcer (of any grade), or bone fracture.
16. Grade 2 or higher peripheral neuropathy.
17. Clinically significant active viral, bacterial or fungal infection
18. Known human immunodeficiency virus seropositivity.
19. Known positive serology for hepatitis B (unless due to vaccination or passive immunization due to immunoglobulin therapy)
20. Known positive serology for hepatitis C (unless due to immunoglobulin therapy)
21. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the trial or evaluation of the trial result
22. History of organ allograft (except for corneal transplant) or autologous or allogeneic bone marrow transplant, or stem cell rescue within 3 months prior to the first dose of IMP
23. Body weight < 40 kg
24. Women who are pregnant or breast feeding.
25. Pulmonary hemorrhage or hemoptysis > 2.5 ml blood within 6 weeks unless cause has been addressed and is medically resolved.
26. History of acute pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2016-11-23 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ignace Vergote, Professor, Principal Investigator — Universitair Ziekenhuizen Leuven
Locations (41):
- United States (20):
  - Mayo Clinic - Phoenix, Phoenix, Arizona
  - University of Colorado Hospital, Aurora, Colorado
  - Yale University, Smilow Cancer Center at Yale New Haven Hospital, New Haven, Connecticut
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University School of Medicine, Winship Cancer Institute, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Belgium (6):
  - Universitair Ziekenhuizen Leuven, Leuven, Flemish Brabant
  - Institut Roi Albert II - Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Brussel - Oncologisch Centrum, Jette
  - Medische oncologie, Oncologisch Centrum - AZ Groeninge, Kortrijk
  - U.Z. Leuven Gasthuisberg, Department of General Medical Oncology, Leuven
  - CHU de Liège, Medical Oncology et. Domaine Universitaire du Sart Tilman, Liège
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark
- Netherlands (4):
  - The Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Leiden University Medical Centre, Leiden
  - Erasmus MC, Medical Oncology, Rotterdam
  - UMC Utrecht Cancer Center, Utrecht
- Spain (6):
  - Hospital Unversitario Vall D'hebron, Barcelona
  - Oncologia Mèdica/ Medical Oncology Department Institut Catalá d'Oncologia (ICO), Barcelona
  - University Hospital of Girona, Girona
  - Hospital Universitario 12 Octubre Servicio de Oncologia Medica, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - University Hospital Lozano Blesa, Aragón Health Research Institute (IIS Aragón), Zaragoza
- United Kingdom (4):
  - University College London Hospitals, London
  - The Christie NHS Foundation Trust Clinical Trials Unit, Manchester
  - Sir Bobby Robson Clinical Trials Unit at the Northern Centre for Cancer Care, Freeman Hospital, Newcastle
  - The Royal Marsden Hospital, Sutton

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W: Participants with relapsed/refractory cancer (ovarian, cervical, endometrial, thyroid, NSCLC, or melanoma) received IV infusion of enapotamab vedotin 0.3 mg/kg 1Q3W until the end of treatment.
- Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W: Participants with relapsed/refractory cancer (ovarian, cervical, endometrial, thyroid, NSCLC, or melanoma) received IV infusion of enapotamab vedotin 0.6 mg/kg 1Q3W until the end of treatment.
- Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W: Participants with relapsed/refractory cancer (ovarian, cervical, endometrial, thyroid, NSCLC, or melanoma) received IV infusion of enapotamab vedotin 1.0 mg/kg 1Q3W until the end of treatment..
- Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W: Participants with relapsed/refractory cancer (ovarian, cervical, endometrial, thyroid, NSCLC, or melanoma) received IV infusion of enapotamab vedotin 1.5 mg/kg 1Q3W until the end of treatment..
- Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W: Participants with relapsed/refractory cancer (ovarian, cervical, endometrial, thyroid, NSCLC, or melanoma) received IV infusion of enapotamab vedotin 2.0 mg/kg 1Q3W until the end of treatment.
- Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W: Participants with relapsed/refractory cancer (ovarian, cervical, endometrial, thyroid, NSCLC, or melanoma) received IV infusion of enapotamab vedotin 2.2 mg/kg 1Q3W until the end of treatment.
- Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W: Participants with relapsed/refractory cancer (ovarian, cervical, endometrial, thyroid, NSCLC, or melanoma) received IV infusion of enapotamab vedotin 2.4 mg/kg 1Q3W until the end of treatment.
- Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W: Participants with relapsed/refractory cancer (ovarian, cervical, endometrial, thyroid, NSCLC, or melanoma) received IV infusion of enapotamab vedotin 0.6 mg/kg 3Q4W until the end of treatment.
- Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W: Participants with relapsed/refractory cancer (ovarian, cervical, endometrial, thyroid, NSCLC, or melanoma) received IV infusion of enapotamab vedotin 0.8 mg/kg 3Q4W until the end of treatment.
- Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W: Participants with relapsed/refractory cancer (ovarian, cervical, endometrial, thyroid, NSCLC, or melanoma) received IV infusion of enapotamab vedotin 1.0 mg/kg 3Q4W until the end of treatment.
- Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W: Participants with relapsed/refractory cancer (ovarian, cervical, endometrial, thyroid, NSCLC, or melanoma) received IV infusion of enapotamab vedotin 1.2 mg/kg 3Q4W until the end of treatment.
- Expansion Part Cohort 1: Enapotamab Vedotin 2.2 mg/kg 1Q3W: Participants with advanced and/or metastatic NSCLC with classical sensitizing epidermal growth factor receptor (EGFR) mutations and/or EGFR mutations targeted by third-generation tyrosine kinase inhibitors, received IV infusion of enapotamab vedotin 2.2 mg/kg 1Q3W until the end of treatment.
- Expansion Part Cohort 3: Enapotamab Vedotin 2.2 mg/kg 1Q3W: Participants with advanced and/or metastatic melanoma with BRAF V600 mutation received IV infusion of enapotamab vedotin 2.2 mg/kg 1Q3W until the end of treatment.
- Expansion Part Cohort 4: Enapotamab Vedotin 2.2 mg/kg 1Q3W: Participants with advanced and/or metastatic melanoma with BRAF V600 wild type received IV infusion of enapotamab vedotin 2.2 mg/kg 1Q3W until the end of treatment.
- Expansion Part Cohort 5: Enapotamab Vedotin 2.2 mg/kg 1Q3W: Participants with advanced and/or metastatic sarcoma received IV infusion of enapotamab vedotin 2.2 mg/kg 1Q3W until the end of treatment.
- Expansion Part Cohort 6: Enapotamab Vedotin 1.0 mg/kg 3Q4W: Participants with advanced and/or metastatic solid tumors (excluding NSCLC, melanoma, sarcoma, and ovarian cancer unless having a known AXL gene amplification) received IV infusion of enapotamab vedotin 1.0 mg/kg 3Q4W until the end of treatment.
- Expansion Part Cohort 7: Enapotamab Vedotin 2.2 mg/kg 1Q3W: Participants with advanced and/or metastatic platinum-resistant ovarian cancer received IV infusion of enapotamab vedotin 2.2 mg/kg 1Q3W until the end of treatment.
- Expansion Part Cohort 2: Enapotamab Vedotin 2.2 mg/kg 1Q3W: Participants with advanced and/or metastatic NSCLC without activating EGFR mutations or anaplastic lymphoma kinase (ALK) rearrangements received IV infusion of enapotamab vedotin 2.2 mg/kg 1Q3W until the end of treatment.
- Expansion Part Cohort 2: Enapotamab Vedotin 1.8 mg/kg 1Q3W: Participants with advanced and/or metastatic NSCLC without activating EGFR mutations or ALK rearrangements received IV infusion of enapotamab vedotin 1.8 mg/kg 1Q3W until the end of treatment.
- Expansion Part Cohort 8: Enapotamab Vedotin 1.0 mg/kg 3Q4W: Participants with advanced and/or metastatic NSCLC without activating EGFR mutations or ALK rearrangements received IV infusion of enapotamab vedotin 1.0 mg/kg 3Q4W until the end of treatment.
Period: Overall Study
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W | Expansion Part Cohort 1: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 3: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 4: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 5: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 6: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Expansion Part Cohort 7: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 1.8 mg/kg 1Q3W | Expansion Part Cohort 8: Enapotamab Vedotin 1.0 mg/kg 3Q4W
Started | 1 | 1 | 3 | 3 | 10 | 11 | 3 | 3 | 3 | 6 | 3 | 22 | 16 | 25 | 25 | 44 | 25 | 55 | 21 | 26
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 3 | 3 | 10 | 11 | 3 | 3 | 3 | 6 | 3 | 22 | 16 | 25 | 25 | 44 | 25 | 55 | 21 | 26
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 3 | 1 | 2 | 1 | 1 | 1 | 1 | 12 | 6 | 6 | 4 | 5 | 4 | 11 | 4 | 2
Not completed — Death | 0 | 1 | 3 | 1 | 6 | 10 | 1 | 2 | 1 | 5 | 1 | 8 | 9 | 17 | 18 | 30 | 17 | 38 | 14 | 16
Not completed — Other | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 3 | 0 | 0
Not completed — Sponsor decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 6 | 2 | 3 | 2 | 7
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set included all participants who received at least 1 dose of enapotamab vedotin. Participants were analyzed according to the assigned treatment/dose (planned dose level and schedule).
Groups:
- Expansion Part Cohort 1: Enapotamab Vedotin 2.2 mg/kg 1Q3W: Participants with advanced and/or classical metastatic NSCLC with classical sensitizing EGFR mutations and/or EGFR mutations targeted by third-generation tyrosine kinase inhibitors) received IV infusion of enapotamab vedotin 2.2 mg/kg 1Q3W until the end of treatment.
- Expansion Part Cohort 2: Enapotamab Vedotin 2.2 mg/kg 1Q3W: Participants with advanced and/or metastatic NSCLC without activating EGFR mutations or ALK rearrangements received IV infusion of enapotamab vedotin 2.2 mg/kg 1Q3W until the end of treatment.
- Total: Total of all reporting groups
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W | Expansion Part Cohort 1: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 3: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 4: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 5: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 6: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Expansion Part Cohort 7: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 1.8 mg/kg 1Q3W | Expansion Part Cohort 8: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Total
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 11 | 3 | 3 | 3 | 6 | 3 | 22 | 16 | 25 | 25 | 44 | 25 | 55 | 21 | 26 | 306
Age, Customized [Count of Participants; unit: Participants]
  >=18 to <65 years | 1 | 0 | 2 | 2 | 9 | 5 | 2 | 1 | 2 | 4 | 3 | 12 | 14 | 13 | 15 | 23 | 16 | 24 | 15 | 17 | 180
  >=65 years | 0 | 1 | 1 | 1 | 1 | 6 | 1 | 2 | 1 | 2 | 0 | 10 | 2 | 12 | 10 | 21 | 9 | 31 | 6 | 9 | 126
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 3 | 7 | 10 | 3 | 2 | 2 | 6 | 3 | 13 | 8 | 7 | 14 | 17 | 25 | 25 | 11 | 13 | 174
  Male | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 1 | 0 | 0 | 9 | 8 | 18 | 11 | 27 | 0 | 30 | 10 | 13 | 132
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 6
  Not Hispanic or Latino | 1 | 1 | 3 | 3 | 10 | 11 | 2 | 3 | 3 | 6 | 3 | 22 | 16 | 24 | 24 | 43 | 23 | 53 | 21 | 25 | 297
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 7
  White | 1 | 1 | 3 | 3 | 10 | 10 | 2 | 3 | 2 | 6 | 3 | 18 | 12 | 21 | 24 | 37 | 20 | 50 | 20 | 23 | 269
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 0 | 1 | 4 | 3 | 0 | 2 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs) for Dose-escalation Part
Description: The DLTs were defined as Grade (G) 4 neutropenia or G4 thrombocytopenia for a minimal duration of 7 days, G3 and G4 febrile neutropenia, >=G3 hemorrhage associated with >=G3 thrombocytopenia, G4 anemia; Stevens Johnson syndrome, toxic epidermal necrolysis, >=G3 cutaneous vasculitis; G3 neuropathy (not improved to G1 within 3 weeks following pausing of dosing) and G4 neuropathy; G3 infusion-related reactions (IRR) that did not resolve to G1 or baseline within 24 hours; G4 IRR or G4 anaphylaxis events; >= G3 diarrhoea and/or vomiting persisting >48 hours or G3 nausea lasting 7 days (both despite optimal medical management); or any >=G3 related non-hematological AEs, which occurred during the Cycle 1 and regarded as medically important as assessed by the Data Monitoring Committee (excluding Grade 3 fatigue or non-hematological laboratory abnormalities as specified in protocol).
Time Frame: From Day 1 to Day 21 of first cycle for 1Q3W dosing regimen and from Day 1 to Day 28 of first cycle for 3Q4W dosing regimen
Population: Dose-determining set included all participants from the Safety Set (participants who received at least 1 dose of enapotamab vedotin, had at least one valid post-baseline safety assessment, and were classified according to first dose received) who either met the minimum exposure criterion and completed the DLT observation period, or who experienced a DLT during Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 10 | 3 | 3 | 3 | 6 | 2
Participants | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 2

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is defined as an AE that meets one of the following criteria: requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, is a congenital anomaly/birth defect, is medically important, results in death, or is life-threatening. In this trial, a TEAE was defined as an AE occurring or worsening between the first dose of enapotamab vedotin and 30 days after the last dose received.
Time Frame: Day 1 through Day 1130 (maximum observed duration)
Population: The safety set included all participants who received at least 1 dose of enapotamab vedotin and had at least one valid post-baseline safety assessment. Participants were classified according to first dose received.
Measure: Count of Participants; unit: Participants
Groups:
- Expansion Part Cohort 1: Enapotamab Vedotin 2.2 mg/kg 1Q3W: Participants with advanced and/or metastatic NSCLC with classical sensitizing EGFR mutations and/or EGFR mutations targeted by third-generation tyrosine kinase inhibitors) received IV infusion of enapotamab vedotin 2.2 mg/kg 1Q3W until the end of treatment.
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W | Expansion Part Cohort 1: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 3: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 4: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 5: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 6: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Expansion Part Cohort 7: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 1.8 mg/kg 1Q3W | Expansion Part Cohort 8: Enapotamab Vedotin 1.0 mg/kg 3Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 11 | 3 | 3 | 3 | 6 | 3 | 22 | 16 | 25 | 25 | 44 | 25 | 56 | 20 | 26
Participants
  Any TEAE | 1 | 1 | 3 | 3 | 10 | 11 | 3 | 3 | 3 | 6 | 3 | 22 | 16 | 25 | 25 | 44 | 25 | 56 | 20 | 26
  Any TESAE | 0 | 0 | 0 | 2 | 7 | 6 | 2 | 1 | 0 | 2 | 3 | 15 | 5 | 16 | 10 | 16 | 12 | 33 | 7 | 14

3. Primary Outcome: Number of Participants With Treatment-emergent Infusion-related AEs and TEAEs Related to Enapotamab Vedotin
Description: Number of participants with treatment-emergent infusion-related AEs and TEAEs related to enapotamab vedotin is reported.
Time Frame: Day 1 through Day 1130 (maximum observed duration)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W | Expansion Part Cohort 1: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 3: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 4: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 5: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 6: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Expansion Part Cohort 7: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 1.8 mg/kg 1Q3W | Expansion Part Cohort 8: Enapotamab Vedotin 1.0 mg/kg 3Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 11 | 3 | 3 | 3 | 6 | 3 | 22 | 16 | 25 | 25 | 44 | 25 | 56 | 20 | 26
Participants
  Treatment emergent infusion-related AEs | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 2 | 1 | 0
  TEAEs related to enapotamab vedotin | 1 | 1 | 3 | 3 | 10 | 10 | 3 | 3 | 3 | 6 | 3 | 21 | 15 | 24 | 24 | 38 | 23 | 52 | 16 | 20

4. Primary Outcome: Number of Participants With >= Grade 3 TEAEs as Assessed by National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.03
Description: Number of participants with TEAEs of >= Grade 3 as assessed by NCI-CTCAE v4.03 is reported. The NCI-CTCAE is a descriptive terminology is used for AE reporting. The NCI-CTCAE v4.03 displays Grades 1 through 5 with unique clinical descriptions of severity for each AE, based on this general guideline: Grade 1 as mild AE, Grade 2 as moderate AE, Grade 3 as severe AE, Grade 4 as life-threatening or disabling AE, and Grade 5 as death. If a participant reported multiple severity grades for an AE, only the maximum grade was used.
Time Frame: Day 1 through Day 1130 (maximum observed duration)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W | Expansion Part Cohort 1: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 3: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 4: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 5: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 6: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Expansion Part Cohort 7: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 1.8 mg/kg 1Q3W | Expansion Part Cohort 8: Enapotamab Vedotin 1.0 mg/kg 3Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 11 | 3 | 3 | 3 | 6 | 3 | 22 | 16 | 25 | 25 | 44 | 25 | 56 | 20 | 26
Participants | 0 | 0 | 0 | 2 | 7 | 9 | 3 | 1 | 0 | 3 | 3 | 15 | 6 | 18 | 16 | 21 | 15 | 40 | 14 | 13

5. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC0-inf) of Conjugated Enapotamab Vedotin for 1Q3W Dose-escalation Part
Description: The AUC0-inf of conjugated enapotamab vedotin for 1Q3W dose-escalation part is reported. Sample scheduling of the 3Q4W dosing regimen did not allow calculation of the specific outcome measure.
Time Frame: Predose, end of infusion (EOI), and 2 and 5 hours after EOI on Day 1 of Cycles 1 and 3
Population: Pharmacokinetic (PK) analysis set included all participants who were exposed to at least 1 dose of enapotamab vedotin and who had at least 1 postdose PK measurement. 'Number analyzed' denotes the number of participants evaluated for the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 11 | 3
day*ug/mL
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 10 | 3
  Cycle 1 Day 1 | 6.143 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 13.233 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 18.353 (8.6) | 40.921 (27.7) | 64.140 (13.2) | 67.998 (32.2) | 76.264 (31.7)
  Cycle 3 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 4 | 0
  Cycle 3 Day 1 | 5.780 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 10.892 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 18.664 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 39.589 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 56.842 (23.8) | 61.161 (10.7) |

6. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Last Measurable Concentration (AUC0-last) of Conjugated Enapotamab Vedotin for 1Q3W Dose-escalation Part
Description: The AUC0-last of conjugated enapotamab vedotin for 1Q3W dose-escalation part is reported. Sample scheduling of the 3Q4W dosing regimen did not allow calculation of the specific outcome measure.
Time Frame: Predose, EOI, and 2 and 5 hours after EOI on Day 1 of Cycles 1 and 3
Population: The PK analysis set included all participants who were exposed to at least 1 dose of enapotamab vedotin and who had at least 1 postdose PK measurement. 'Number analyzed' denotes the number of participants evaluated for the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 11 | 3
day*ug/mL
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 10 | 3
  Cycle 1 Day 1 | 5.509 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 10.369 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 16.004 (18.5) | 36.526 (29.7) | 58.410 (11.6) | 62.563 (29.7) | 71.196 (32.5)
  Cycle 3 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 4 | 0
  Cycle 3 Day 1 | 5.306 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 9.157 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 15.047 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 36.333 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 51.541 (21.4) | 57.759 (11.9) |

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Conjugated Enapotamab Vedotin for Dose-escalation Part
Description: The Cmax of conjugated enapotamab vedotin for dose-escalation part is reported.
Time Frame: For 1Q3W dosing regimen: Predose, EOI, and 2 and 5 hours after EOI on Day 1 of Cycles 1 and 3; For 3Q4W dosing regimen: Predose and EOI on Days 1 and 8 of Cycles 1 and 3; and predose, EOI, and 2 and 5 hours after EOI on Day 15 of Cycles 1 and 3
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 11 | 3 | 3 | 3 | 6 | 3
ug/mL
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 10 | 3 | 3 | 2 | 6 | 3
  Cycle 1 Day 1 | 7.250 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 12.600 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 16.615 (16.7) | 33.005 (9.4) | 39.647 (11.4) | 43.377 (25.6) | 48.548 (33.0) | 10.127 (40.2) | 14.307 (31.6) | 18.040 (12.0) | 17.928 (22.0)
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 6 | 3
  Cycle 1 Day 8 |  |  |  |  |  |  |  | 14.201 (11.9) | 16.765 (36.3) | 18.698 (8.1) | 18.958 (19.5)
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 6 | 1
  Cycle 1 Day 15 |  |  |  |  |  |  |  | 13.172 (8.0) | 16.166 (37.2) | 16.991 (7.8) | 18.500 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm.
  Cycle 3 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 4 | 0 | 0 | 1 | 1 | 0
  Cycle 3 Day 1 | 6.870 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 11.000 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 16.200 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 32.400 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 35.890 (17.9) | 38.928 (9.0) |  |  | 22.400 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 21.800 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. |
  Cycle 3 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Cycle 3 Day 8 |  |  |  |  |  |  |  |  | 21.200 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. |  |
  Cycle 3 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Cycle 3 Day 15 |  |  |  |  |  |  |  |  | 24.100 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 22.800 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. |

8. Secondary Outcome: Total Clearance (CL) of Conjugated Enapotamab Vedotin in Dose-escalation Part
Description: The total CL of conjugated enapotamab vedotin in dose-escalation part is reported.
Time Frame: For 1Q3W dosing regimen: Predose, EOI, and 2 and 5 hours after EOI on Day 1 of Cycles 1 and 3; For 3Q4W dosing regimen: EOI, and 2 and 5 hours after EOI on Day 15 of Cycles 1 and 3
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 11 | 3 | 3 | 3 | 6 | 3
L/day
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 10 | 3 | 0 | 0 | 0 | 0
  Cycle 1 Day 1 | 4.053 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 3.446 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 3.538 (21.8) | 2.307 (28.3) | 2.202 (22.2) | 2.205 (25.4) | 1.783 (24.3) |  |  |  |
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 6 | 1
  Cycle 1 Day 15 |  |  |  |  |  |  |  | 3.679 (9.4) | 3.084 (93.8) | 3.402 (31.3) | 2.629 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm.
  Cycle 3 day 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 4 | 0 | 0 | 0 | 0 | 0
  Cycle 3 day 1 | 4.360 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 4.187 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 3.000 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 2.160 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 2.285 (27.1) | 2.539 (14.7) |  |  |  |  |
  Cycle 3 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Cycle 3 Day 15 |  |  |  |  |  |  |  |  | 2.281 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 3.412 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. |

9. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax) of Conjugated Enapotamab Vedotin for Dose-escalation Part
Description: The Tmax of conjugated enapotamab vedotin for dose-escalation part is reported.
Time Frame: For 1Q3W dosing regimen: Predose, EOI, and 2 and 5 hours after EOI on Day 1 of Cycles 1 and 3; For 3Q4W dosing regimen: Predose, EOI, and 2 and 5 hours after EOI on Day 15 of Cycles 1 and 3
Population: as for outcome 6
Measure: Median (Full Range); unit: Day
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 11 | 3 | 3 | 3 | 6 | 3
Day
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 10 | 3 | 0 | 0 | 0 | 0
  Cycle 1 Day 1 | 0.06 [0.06 to 0.06] | 0.03 [0.03 to 0.03] | 0.036 [0.03 to 0.04] | 0.033 [0.03 to 0.04] | 0.032 [0.02 to 0.09] | 0.032 [0.02 to 0.04] | 0.03 [0.02 to 0.03] |  |  |  |
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 6 | 1
  Cycle 1 Day 15 |  |  |  |  |  |  |  | 14.010 [13.96 to 14.88] | 14.058 [13.98 to 14.08] | 14.083 [14.00 to 14.19] | 13.98 [13.98 to 13.98]
  Cycle 3 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 4 | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1 | 0.04 [0.04 to 0.04] | 0.03 [0.03 to 0.03] | 0.04 [0.04 to 0.04] | 0.030 [0.03 to 0.03] | 0.036 [0.02 to 0.05] | 0.042 [0.03 to 0.11] |  |  |  |  |
  Cycle 3 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Cycle 3 Day 15 |  |  |  |  |  |  |  |  | 14.02 [14.02 to 14.02] | 13.98 [13.98 to 13.98] |

10. Secondary Outcome: Half-life Lambda-z (t1/2) of Conjugated Enapotamab Vedotin for Dose-escalation Part
Description: The t1/2 of conjugated enapotamab vedotin for dose-escalation part is reported.
Time Frame: as for outcome 9
Population: as for outcome 6
Measure: Median (Full Range); unit: Day
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 11 | 3 | 3 | 3 | 6 | 3
Day
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 10 | 3 | 0 | 0 | 0 | 0
  Cycle 1 Day 1 | 0.87 [0.87 to 0.87] | 1.49 [1.49 to 1.49] | 1.362 [1.02 to 1.39] | 1.384 [1.19 to 1.65] | 2.004 [1.67 to 2.53] | 1.810 [1.53 to 2.74] | 2.153 [1.99 to 2.60] |  |  |  |
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 6 | 1
  Cycle 1 Day 15 |  |  |  |  |  |  |  | 1.097 [0.66 to 1.56] | 1.398 [0.91 to 1.81] | 1.423 [0.77 to 1.96] | 2.05 [2.05 to 2.05]
  Cycle 3 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 4 | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1 | 0.78 [0.78 to 0.78] | 1.07 [1.07 to 1.07] | 1.130 [1.13 to 1.13] | 1.68 [1.68 to 1.68] | 2.117 [1.55 to 2.90] | 2.035 [1.38 to 2.74] |  |  |  |  |
  Cycle 3 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Cycle 3 Day 15 |  |  |  |  |  |  |  |  | 1.51 [1.51 to 1.51] | 1.44 [1.44 to 1.44] |

11. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Conjugated Enapotamab Vedotin for Dose-escalation Part
Description: The Vss of conjugated enapotamab vedotin for dose-escalation part is reported.
Time Frame: as for outcome 9
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 11 | 3 | 3 | 3 | 6 | 3
L/day
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 10 | 3 | 0 | 0 | 0 | 0
  Cycle 1 Day 1 | 4.909 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 6.544 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 5.873 (9.8) | 4.208 (12.5) | 6.028 (18.4) | 5.489 (24.2) | 5.038 (27.3) |  |  |  |
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 6 | 1
  Cycle 1 Day 15 |  |  |  |  |  |  |  | 57.736 (10.0) | 48.001 (91.1) | 53.436 (28.0) | 42.708 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm.
  Cycle 3 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 4 | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1 | 4.755 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 6.288 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 4.870 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 4.534 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 6.072 (24.2) | 6.656 (22.0) |  |  |  |  |
  Cycle 3 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Cycle 3 Day 15 |  |  |  |  |  |  |  |  | 36.476 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 53.085 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. |

12. Secondary Outcome: AUC0-inf of Free Toxin Monomethyl Auristatin E (MMAE) for 1Q3W Dose-escalation Part
Description: The AUC0-inf of MMAE for 1Q3W dose-escalation part is reported. Sample scheduling of the 3Q4W dosing regimen did not allow calculation of the specific outcome measure.
Time Frame: Predose, EOI, and 2 and 5 hours after EOI on Day 1 of Cycles 1 and 3
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*pg/mL
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 11 | 3
day*pg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 10 | 2
  Cycle 1 Day 1 | 3832.48 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 6144.11 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 13673.7 (110.4) | 26549.1 (82.9) | 33494.5 (47.1) | 50459.6 (117.0) | 48626.4 (95.5)
  Cycle 3 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 4 | 1
  Cycle 3 Day 1 | 3248.46 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 7452.05 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 4338.20 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 47093.9 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 30512.0 (47.8) | 34188.6 (46.6) | 16754.5 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm.

13. Secondary Outcome: AUC0-last of MMAE for 1Q3W Dose-escalation Part
Description: The AUC0-last of MMAE for 1Q3W dose-escalation part is reported. Sample scheduling of the 3Q4W dosing regimen did not allow calculation of the specific outcome measure.
Time Frame: Predose, EOI, and 2 and 5 hours after EOI on Day 1 of Cycles 1 and 3
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*pg/mL
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 11 | 3
day*pg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 10 | 3
  Cycle 1 Day 1 | 3364.64 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 5980.86 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 13194.4 (110.4) | 25549.3 (80.8) | 31854.7 (46.4) | 34659.4 (81.2) | 38963.5 (65.4)
  Cycle3 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 4 | 1
  Cycle3 Day 1 | 2642.23 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 7263.16 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 4156.66 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 44553.3 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 28890.0 (47.4) | 31429.9 (43.2) | 16354.3 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm.

14. Secondary Outcome: Cmax of MMAE for Dose-escalation Part
Description: The Cmax of MMAE for dose-escalation part is reported.
Time Frame: as for outcome 7
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 11 | 3 | 3 | 3 | 6 | 3
pg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 10 | 3 | 3 | 3 | 6 | 3
  Cycle 1 Day 1 | 700.000 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 947.000 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 1874.13 (5) | 4036.47 (81.8) | 4265.60 (46.1) | 5154.58 (61.9) | 5617.89 (34.7) | 161.140 (75.0) | 175.315 (159.4) | 303.977 (45.3) | 244.623 (48.9)
  Cycle 1 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 6 | 3
  Cycle 1 Day 8 |  |  |  |  |  |  |  | 738.227 (28.2) | 766.467 (91.4) | 1982.67 (58.1) | 1553.93 (86.2)
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 6 | 1
  Cycle 1 Day 15 |  |  |  |  |  |  |  | 1715.54 (42.8) | 2525.75 (54.7) | 4379.50 (58.2) | 3720.00 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm.
  Cycle 3 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 4 | 1 | 0 | 1 | 1 | 0
  Cycle 3 Day 1 | 631.000 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 1200.000 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 628.000 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 6500.00 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 3964.40 (49.4) | 4127.31 (39.3) | 2180.00 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. |  | 442.000 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 558.000 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. |
  Cycle 3 Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Cycle 3 Day 8 |  |  |  |  |  |  |  |  | 1060.00 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. |  |
  Cycle 3 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Cycle 3 Day 15 |  |  |  |  |  |  |  |  | 2960.00 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 5190.00 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. |

15. Secondary Outcome: Total CL of MMAE in Dose-escalation Part
Description: The total CL of MMAE in dose-escalation part is reported.
Time Frame: as for outcome 8
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 11 | 3 | 3 | 3 | 6 | 3
L/day
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 10 | 2 | 0 | 0 | 0 | 0
  Cycle 1 Day 1 | 6497.09 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 7421.74 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 4748.64 (87.2) | 3555.78 (90.6) | 4216.71 (42.0) | 2971.09 (107.2) | 2813.05 (35.9) |  |  |  |
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 6 | 0
  Cycle 1 Day 15 |  |  |  |  |  |  |  | 4819.44 (25.8) | 4666.23 (35.5) | 2847.55 (46.7) |
  Cycle 3 day 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 4 | 1 | 0 | 0 | 0 | 0
  Cycle 3 day 1 | 7757.51 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 6119.12 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 12908.6 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 1815.52 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 4256.44 (50.1) | 4542.22 (42.8) | 5849.18 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. |  |  |  |
  Cycle 3 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Cycle 3 Day 15 |  |  |  |  |  |  |  |  | 3899.39 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. | 2507.90 (NA) — Geometric coefficient of variation was not derived as only one participant was evaluated for this arm. |

16. Secondary Outcome: Tmax of MMAE for Dose-escalation Part
Description: The Tmax of MMAE for dose-escalation part is reported.
Time Frame: as for outcome 9
Population: as for outcome 6
Measure: Median (Full Range); unit: Day
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 11 | 3 | 3 | 3 | 6 | 3
Day
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 10 | 3 | 0 | 0 | 0 | 0
  Cycle 1 Day 1 | 2.95 [2.95 to 2.95] | 3.00 [3.00 to 3.00] | 2.938 [2.89 to 2.94] | 2.764 [2.72 to 2.83] | 2.852 [0.97 to 3.03] | 2.866 [1.00 to 6.85] | 2.942 [2.82 to 7.00] |  |  |  |
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 6 | 1
  Cycle 1 Day 15 |  |  |  |  |  |  |  | 15.950 [15.93 to 17.73] | 15.982 [15.97 to 15.99] | 15.911 [14.51 to 15.95] | 20.820 [20.82 to 20.82]
  Cycle 3 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 4 | 1 | 0 | 0 | 0 | 0
  Cycle 3 Day 1 | 2.83 [2.83 to 2.83] | 2.87 [2.87 to 2.87] | 0.94 [0.94 to 0.94] | 2.83 [2.83 to 2.83] | 2.830 [0.94 to 3.96] | 2.727 [0.94 to 2.94] | 3.02 [3.02 to 3.02] |  |  |  |
  Cycle 3 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Cycle 3 Day 15 |  |  |  |  |  |  |  |  | 14.93 [14.93 to 14.93] | 15.890 [15.89 to 15.89] |

17. Secondary Outcome: t1/2 of MMAE for Dose-escalation Part
Description: The t1/2 of MMAE for dose-escalation part is reported.
Time Frame: as for outcome 9
Population: as for outcome 6
Measure: Median (Full Range); unit: Day
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 11 | 3 | 3 | 3 | 6 | 3
Day
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 10 | 2 | 0 | 0 | 0 | 0
  Cycle 1 Day 1 | 2.19 [2.19 to 2.19] | 2.35 [2.35 to 2.35] | 2.470 [2.10 to 2.70] | 2.620 [1.85 to 2.98] | 2.420 [2.02 to 3.75] | 3.128 [1.55 to 42.73] | 2.835 [2.45 to 3.22] |  |  |  |
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 6 | 0
  Cycle 1 Day 15 |  |  |  |  |  |  |  | 3.976 [2.78 to 6.06] | 3.115 [2.49 to 5.04] | 4.739 [2.85 to 8.70] |
  Cycle 3 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 4 | 1 | 0 | 0 | 0 | 0
  Cycle 3 Day 1 | 1.94 [1.94 to 1.94] | 2.32 [2.32 to 2.32] | 2.71 [2.71 to 2.71] | 2.52 [2.52 to 2.52] | 2.746 [2.18 to 3.12] | 3.364 [2.85 to 4.99] | 1.98 [1.98 to 1.98] |  |  |  |
  Cycle 3 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Cycle 3 Day 15 |  |  |  |  |  |  |  |  | 2.330 [2.33 to 2.33] | 3.37 [3.37 to 3.37] |

18. Secondary Outcome: Number of Participants With Antidrug Antibodies (ADAs) Confirmed Positive to Enapotamab Vedotin
Description: The ADA assessment was performed according to a tiered approach. First samples were screened for an ADA response; positively screened samples were analyzed in a confirmation method. Subsequently confirmed positive samples were analyzed for titre and the presence of neutralizing antibodies. Number of participants with ADA confirmed positive to enapotamab vedotin is reported.
Time Frame: Day 1 through Day 1130 (Dose-escalation part: Predose of Day 1 of Cycles 1 to 12, end of treatment [EOT], and 30 days after last study drug; Expansion part: Predose on Day 1 of Cycles 1 to 5, then every fourth cycle until PD)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W | Expansion Part Cohort 1: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 3: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 4: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 5: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 6: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Expansion Part Cohort 7: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 1.8 mg/kg 1Q3W | Expansion Part Cohort 8: Enapotamab Vedotin 1.0 mg/kg 3Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 11 | 3 | 3 | 3 | 6 | 3 | 22 | 16 | 25 | 25 | 44 | 25 | 56 | 20 | 26
Participants | 0 | 0 | 1 | 1 | 5 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 4 | 1 | 3 | 0 | 7 | 5 | 0 | 0

19. Secondary Outcome: Number of Participants With Objective Response (OR) Based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) As Assessed by Investigator
Description: Radiological evaluation based on RECIST v1.1 was performed by the investigator using computed tomography (CT) scans/ magnetic resonance imaging (MRI) scans/ positron emission tomography (PET) scans. The OR was defined as confirmed CR or confirmed PR per RECIST v1.1. The changes in tumor measurements that were confirmed by repeat assessments performed no less than 4 weeks after initial response are called confirmed responses. The CR was defined as disappearance of all target and non-target lesions and all pathological lymph nodes must have decreased to < 10 mm in short axis. The PR was defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions taking as reference the baseline sum of LD.
Time Frame: Day 1 through 44.5 months (maximum observed duration)
Population: The full analysis set included all participants who received at least 1 dose of enapotamab vedotin. Participants were classified according to first dose received.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W | Expansion Part Cohort 1: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 3: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 4: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 5: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 6: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Expansion Part Cohort 7: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 1.8 mg/kg 1Q3W | Expansion Part Cohort 8: Enapotamab Vedotin 1.0 mg/kg 3Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 11 | 3 | 3 | 3 | 6 | 3 | 22 | 16 | 25 | 25 | 44 | 25 | 55 | 21 | 26
Participants | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 4 | 2 | 5 | 1 | 3

20. Secondary Outcome: Number of Participants With Best Cancer Antigen 125 (CA-125) Response
Description: The best CA-125 response was evaluated in participants with ovarian cancer. A CA-125 partial response was defined as at least a 50% reduction in CA-125 levels in blood from a pretreatment sample. Participants who had a CA-125 partial response and had CA-125 level falls to within the reference range (0-35 units/mL) were classified as CA-125 complete responders. The response was confirmed and maintained for at least 28 days. The best overall response (CA-125 partial response and CA-125 complete response) is reported.
Time Frame: From Screening (within 2 weeks before starting of the study treatment) through Day 1130 (maximum observed duration)
Population: Participants from the full analysis set with ovarian cancer who had an initial CA-125 level of at least twice the upper limit of the reference range within 2 weeks before starting the study treatment were evaluated for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W | Expansion Part Cohort 1: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 3: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 4: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 5: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 6: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Expansion Part Cohort 7: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 1.8 mg/kg 1Q3W | Expansion Part Cohort 8: Enapotamab Vedotin 1.0 mg/kg 3Q4W
Number analyzed (Participants) | 0 | 1 | 0 | 1 | 3 | 3 | 1 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 19 | 0 | 0 | 0
Participants
  CA-125 partial response |  | 0 |  | 0 | 0 | 0 | 1 | 0 |  | 0 | 0 |  |  |  |  |  | 2 |  |  |
  CA-125 complete response |  | 0 |  | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 |  |  |  |  |  | 0 |  |  |

21. Secondary Outcome: Duration of Response (DoR) Based on RECIST v1.1 as Assessed by Investigator for Expansion Part
Description: The DoR was defined as the number of months from the first documentation of objective tumor response (CR or PR) to the date of first progressive disease (PD) or death. The OR was defined as confirmed CR or confirmed PR per RECIST v1.1. The changes in tumor measurements that were confirmed by repeat assessments performed no less than 4 weeks after initial response are called confirmed responses. The CR was defined as disappearance of all target and non-target lesions and all pathological lymph nodes must have decreased to < 10 mm in short axis. The PR was defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions taking as reference the baseline sum of LD. The PD was defined as at least 20% increase in the sum of LD of target lesions taking as reference the smallest sum of the LD recorded since the treatment started or the appearance of one or more new target and non-target lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Day 1 through 44.5 months (maximum observed duration)
Population: The full analysis set included all participants who received at least 1 dose of enapotamab vedotin. Participants were classified according to first dose received. Participants who achieved confirmed OR by the investigator assessment were evaluated for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Expansion Part Cohort 1: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 3: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 4: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 5: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 6: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Expansion Part Cohort 7: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 1.8 mg/kg 1Q3W | Expansion Part Cohort 8: Enapotamab Vedotin 1.0 mg/kg 3Q4W
Number analyzed (Participants) | 0 | 1 | 2 | 0 | 2 | 1 | 1 | 1 | 1
Months |  | 4.2 [NA to NA] — 95% confidence interval was not reached due to an insufficient events being observed. | 4.1 [2.4 to NA] — Upper limit of 95% confidence interval was not reached due to an insufficient events being observed. |  | 4.9 [2.6 to NA] — Upper limit of 95% confidence interval was not reached due to an insufficient events being observed. | 3.0 [NA to NA] — 95% confidence interval was not reached due to an insufficient events being observed. | NA [3.0 to NA] — Median and upper limit of 95% confidence interval was not reached due to an insufficient events being observed. | 3.0 [NA to NA] — 95% confidence interval was not reached due to an insufficient events being observed. | 4.9 [NA to NA] — 95% confidence interval was not reached due to an insufficient events being observed.

22. Secondary Outcome: Progression Free Survival (PFS) as Assessed by Investigator
Description: The PFS was defined as the number of months from the date of first study drug administration to first PD or death. The PD was defined as at least 20% increase in the sum of longest diameters of target lesions taking as reference the smallest sum of the longest diameters recorded since the treatment started or the appearance of one or more new lesions. The PFS was estimated using Kaplan-Meier method.
Time Frame: Day 1 through 44.5 months (maximum observed duration)
Population: as for outcome 19
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Expansion Part Cohort 7: Enapotamab Vedotin 2.2 mg/kg 1Q3W; Expansion Part Cohort 2: Enapotamab Vedotin 2.2 mg/kg 1Q3W: Participants with advanced and/or metastatic NSCLC without activating EGFR mutations or ALK rearrangements received IV infusion of enapotamab vedotin 2.2 mg/kg 1Q3W until the end of treatment.
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W | Expansion Part Cohort 1: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 3: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 4: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 5: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 6: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Expansion Part Cohort 7: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 1.8 mg/kg 1Q3W | Expansion Part Cohort 8: Enapotamab Vedotin 1.0 mg/kg 3Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 11 | 3 | 3 | 3 | 6 | 3 | 22 | 16 | 25 | 25 | 44 | 25 | 55 | 21 | 26
Months | 6.7 [NA to NA] — 95% confidence interval was not reached due to an insufficient events being observed. | 3.5 [NA to NA] — 95% confidence interval was not reached due to an insufficient events being observed. | 1.3 [1.2 to NA] — Upper limit of 95% confidence interval was not reached due to an insufficient events being observed. | 5.3 [1.1 to NA] — Upper limit of 95% confidence interval was not reached due to an insufficient events being observed. | 2.8 [1.4 to NA] — Upper limit of 95% confidence interval was not reached due to an insufficient events being observed. | 2.6 [0.7 to NA] — Upper limit of 95% confidence interval was not reached due to an insufficient events being observed. | NA [NA to NA] — Median and 95% confidence interval were not reached due to an insufficient events being observed. | 1.6 [NA to NA] — 95% confidence interval was not reached due to an insufficient events being observed. | 1.6 [1.3 to NA] — Upper limit of 95% confidence interval was not reached due to an insufficient events being observed. | 4.3 [1.0 to NA] — Upper limit of 95% confidence interval was not reached due to an insufficient events being observed. | 0.8 [0.4 to NA] — Upper limit of 95% confidence interval was not reached due to an insufficient events being observed. | 2.6 [1.2 to 2.8] | 2.6 [1.2 to 3.9] | 2.8 [1.3 to 5.0] | 2.6 [1.4 to 4.1] | 1.9 [1.6 to 2.1] | 1.6 [1.3 to 3.0] | 2.2 [1.4 to 3.9] | 2.6 [1.1 to 4.0] | 2.0 [1.4 to 4.1]

23. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the number of months from date of first study drug administration to death. The OS was estimated using Kaplan-Meier method.
Time Frame: Day 1 through 44.5 months (maximum observed duration)
Population: as for outcome 19
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Expansion Part Cohort 5: Enapotamab Vedotin 2.2 mg/kg 1Q3W: Participants with advanced and/or metastatic sarcoma received IV infusion of enapotamab vedotin 2.2 mg/kg 1Q3W until the end of treatment.st.
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W | Expansion Part Cohort 1: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 3: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 4: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 5: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 6: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Expansion Part Cohort 7: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 1.8 mg/kg 1Q3W | Expansion Part Cohort 8: Enapotamab Vedotin 1.0 mg/kg 3Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 11 | 3 | 3 | 3 | 6 | 3 | 22 | 16 | 25 | 25 | 44 | 25 | 55 | 21 | 26
Months | NA [NA to NA] — Median and 95% confidence interval were not reached due to an insufficient events being observed. | 4.3 [NA to NA] — 95% confidence interval was not reached due to an insufficient events being observed. | 6.4 [6.3 to NA] — Upper limit of 95% confidence interval was not reached due to an insufficient events being observed. | NA [6.7 to NA] — Median and upper limit of 95% confidence interval were not reached due to an insufficient events being observed. | 14.5 [3.1 to NA] — Upper limit of 95% confidence interval was not reached due to an insufficient events being observed. | 7.6 [2.2 to 12.1] | 44.5 [NA to NA] — 95% confidence interval was not reached due to an insufficient events being observed. | 6.7 [6.7 to NA] — Upper limit of 95% confidence interval was not reached due to an insufficient events being observed. | 14.3 [NA to NA] — 95% confidence interval was not reached due to an insufficient events being observed. | 7.7 [4.3 to NA] — Upper limit of 95% confidence interval was not reached due to an insufficient events being observed. | 21.7 [0.4 to NA] — Upper limit of 95% confidence interval was not reached due to an insufficient events being observed. | 16.5 [4.1 to 25.9] | 8.6 [3.6 to 19.1] | 9.2 [4.0 to 14.9] | 17.1 [5.7 to 24.3] | 7.0 [5.2 to 11.6] | 8.4 [6.5 to 12.4] | 11.3 [8.0 to 15.5] | 8.7 [5.8 to 14.1] | 8.0 [4.1 to 12.9]

24. Secondary Outcome: Change in AXL Expression (Total Tumor H-score) From Baseline to EOT Visit for Expansion Part
Description: Change in AXL expression (total humor H-score in membrane or cytoplasm) from Baseline to EOT visit for the expansion part is reported. The H-score captures both the intensity and proportion of AXL positive tumor cells and was defined by the formula: H-score = (1 × % 1+ tumor cells) + (2 × % 2+ tumor cells) + (3 × % 3+ tumor cells); where '1+' indicates weak staining intensity, '2+' indicates medium staining intensity, and '3+' indicates strong staining intensity. The H-score values ranges from 0 to 300. Lower H-scores represent lower AXL expression in the tumor sample, while higher scores represent stronger AXL expression in the tumor samples.
Time Frame: Baseline (Study Days -21 to 1) and EOT visit (Day 1100)
Population: The full analysis set included all participants who received at least 1 dose of enapotamab vedotin. Participants were classified according to first dose received in the expansion part. Participants who had tumor H-scores in membrane or cytoplasm assessed at Baseline and at the end of treatment visit were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Expansion Part Cohort 1: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 3: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 4: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 5: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 6: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Expansion Part Cohort 7: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 1.8 mg/kg 1Q3W | Expansion Part Cohort 8: Enapotamab Vedotin 1.0 mg/kg 3Q4W
Number analyzed (Participants) | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Score on a scale | -8.0 (NA) — Standard deviation was not derived as only one participant was evaluated. | -1.0 (NA) — Standard deviation was not derived as only one participant was evaluated. |  | -30.0 (NA) — Standard deviation was not derived as only one participant was evaluated. |  | 35.0 (NA) — Standard deviation was not derived as only one participant was evaluated. | -14.0 (NA) — Standard deviation was not derived as only one participant was evaluated. |  |

25. Primary Outcome: Number of Participants With Grade 3 or 4 Laboratory Results
Description: Number of participants with laboratory measurements graded as Grade 3 or 4 by NCI-CTCAE v 4.03 is reported.
Time Frame: Day 1 through Day 1130 (maximum observed duration)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W | Expansion Part Cohort 1: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 3: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 4: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 5: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 6: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Expansion Part Cohort 7: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 1.8 mg/kg 1Q3W | Expansion Part Cohort 8: Enapotamab Vedotin 1.0 mg/kg 3Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 10 | 11 | 3 | 3 | 3 | 6 | 3 | 22 | 16 | 25 | 25 | 44 | 25 | 56 | 20 | 26
Participants
  Activated partial thromboplastin time | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
  Alanine aminotransferase | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1
  Amylase | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 1
  Aspartate aminotransferase | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0
  Calcium | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Gamma-glutamyl transferase | 0 | 1 | 0 | 0 | 1 | 4 | 1 | 0 | 1 | 1 | 2 | 5 | 0 | 3 | 0 | 7 | 4 | 8 | 1 | 3
  Leukocytes | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 1 | 2 | 2 | 1
  Lipase | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 1 | 2 | 1 | 1 | 3 | 4 | 3 | 1
  Lymphocytes | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 2 | 0 | 5 | 0 | 5 | 7 | 9 | 8 | 9 | 2 | 4
  Magnesium | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Neutrophils | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 7 | 3 | 5 | 8 | 2 | 2
  Potassium | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1
  Prothrombin Intl. Normalized Ratio | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 4 | 0 | 1
  Sodium | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 4 | 2 | 3 | 7 | 1 | 3
  Triglycerides | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 2 | 3 | 1 | 1 | 1 | 0 | 0
  Alkaline Phosphatase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1
  Hemoglobin | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 3 | 1 | 2 | 0 | 0
  Albumin | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Bilirubin | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Cholesterol | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: For TEAEs: Day 1 through Day 1130 and for all-cause mortality: From date of inform consent form until death (up to 44.5 months) (maximum observed duration)
Description: The TEAEs were evaluated per the safety set and all-cause mortality was evaluated per the full analysis set.
Groups:
- Expansion Part Cohort 1: Enapotamab Vedotin 2.2 mg/kg 1Q3W: Participants with advanced and/or metastatic NSCLC with classical sensitizing classical EGFR mutations and/or EGFR mutations targeted by third-generation tyrosine kinase inhibitors) received IV infusion of enapotamab vedotin 2.2 mg/kg 1Q3W until the end of treatment.
Arm/Group | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W | Expansion Part Cohort 1: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 3: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 4: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 5: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 6: Enapotamab Vedotin 1.0 mg/kg 3Q4W | Expansion Part Cohort 7: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 2.2 mg/kg 1Q3W | Expansion Part Cohort 2: Enapotamab Vedotin 1.8 mg/kg 1Q3W | Expansion Part Cohort 8: Enapotamab Vedotin 1.0 mg/kg 3Q4W
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/1 | 3/3 | 1/3 | 6/10 | 10/11 | 1/3 | 2/3 | 1/3 | 5/6 | 1/3 | 8/22 | 9/16 | 17/25 | 18/25 | 30/44 | 17/25 | 38/56 | 14/22 | 16/26
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/3 | 2/3 | 7/10 | 6/11 | 2/3 | 1/3 | 0/3 | 2/6 | 3/3 | 15/22 | 5/16 | 16/25 | 10/25 | 16/44 | 12/25 | 33/56 | 7/20 | 14/26
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 3/3 | 3/3 | 10/10 | 11/11 | 3/3 | 3/3 | 3/3 | 6/6 | 3/3 | 22/22 | 16/16 | 24/25 | 25/25 | 44/44 | 25/25 | 56/56 | 20/20 | 23/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W (N=1) | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W (N=1) | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W (N=3) | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W (N=3) | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W (N=10) | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W (N=11) | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W (N=3) | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W (N=3) | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W (N=3) | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W (N=6) | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W (N=3) | Expansion Part Cohort 1: Enapotamab Vedotin 2.2 mg/kg 1Q3W (N=22) | Expansion Part Cohort 3: Enapotamab Vedotin 2.2 mg/kg 1Q3W (N=16) | Expansion Part Cohort 4: Enapotamab Vedotin 2.2 mg/kg 1Q3W (N=25) | Expansion Part Cohort 5: Enapotamab Vedotin 2.2 mg/kg 1Q3W (N=25) | Expansion Part Cohort 6: Enapotamab Vedotin 1.0 mg/kg 3Q4W (N=44) | Expansion Part Cohort 7: Enapotamab Vedotin 2.2 mg/kg 1Q3W (N=25) | Expansion Part Cohort 2: Enapotamab Vedotin 2.2 mg/kg 1Q3W (N=56) | Expansion Part Cohort 2: Enapotamab Vedotin 1.8 mg/kg 1Q3W (N=20) | Expansion Part Cohort 8: Enapotamab Vedotin 1.0 mg/kg 3Q4W (N=26)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac Tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 7 (7) | 4 (4) | 4 (4) | 3 (3) | 2 (2) | 0 (0) | 3 (4) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
General Physical Health Deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Influenza Like Illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple Organ Dysfunction Syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary Obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Portal Vein Thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis Infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neutropenic Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis Jirovecii Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Staphylococcal Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphangiosis Carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to Peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial Effusion Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Motor-Sensory Axonal Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss Of Consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Monoplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Partial Seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral Motor Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral Sensorimotor Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device Occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Tracheal Obstruction Extrinsic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose-escalation Part: Enapotamab Vedotin 0.3 mg/kg 1Q3W (N=1) | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 1Q3W (N=1) | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 1Q3W (N=3) | Dose-escalation Part: Enapotamab Vedotin 1.5 mg/kg 1Q3W (N=3) | Dose-escalation Part: Enapotamab Vedotin 2.0 mg/kg 1Q3W (N=10) | Dose-escalation Part: Enapotamab Vedotin 2.2 mg/kg 1Q3W (N=11) | Dose-escalation Part: Enapotamab Vedotin 2.4 mg/kg 1Q3W (N=3) | Dose-escalation Part: Enapotamab Vedotin 0.6 mg/kg 3Q4W (N=3) | Dose-escalation Part: Enapotamab Vedotin 0.8 mg/kg 3Q4W (N=3) | Dose-escalation Part: Enapotamab Vedotin 1.0 mg/kg 3Q4W (N=6) | Dose-escalation Part: Enapotamab Vedotin 1.2 mg/kg 3Q4W (N=3) | Expansion Part Cohort 1: Enapotamab Vedotin 2.2 mg/kg 1Q3W (N=22) | Expansion Part Cohort 3: Enapotamab Vedotin 2.2 mg/kg 1Q3W (N=16) | Expansion Part Cohort 4: Enapotamab Vedotin 2.2 mg/kg 1Q3W (N=25) | Expansion Part Cohort 5: Enapotamab Vedotin 2.2 mg/kg 1Q3W (N=25) | Expansion Part Cohort 6: Enapotamab Vedotin 1.0 mg/kg 3Q4W (N=44) | Expansion Part Cohort 7: Enapotamab Vedotin 2.2 mg/kg 1Q3W (N=25) | Expansion Part Cohort 2: Enapotamab Vedotin 2.2 mg/kg 1Q3W (N=56) | Expansion Part Cohort 2: Enapotamab Vedotin 1.8 mg/kg 1Q3W (N=20) | Expansion Part Cohort 8: Enapotamab Vedotin 1.0 mg/kg 3Q4W (N=26)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 4 (8) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 3 (10) | 0 (0) | 4 (6) | 2 (2) | 3 (6) | 4 (6) | 6 (8) | 3 (3) | 11 (14) | 3 (3) | 4 (5)
Anaemia Macrocytic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (9) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (4) | 4 (29) | 2 (3) | 2 (6) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 3 (6) | 2 (2) | 5 (11) | 7 (13) | 2 (3) | 9 (14) | 7 (9) | 3 (5) | 0 (0)
Normocytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (4) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 2 (2)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Borderline Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival Haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry Eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (2) | 1 (3) | 0 (0)
Eye Irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye Pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacrimation Increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular Hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trichomegaly (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Visual Impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous Floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 4 (7) | 2 (4) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 4 (7) | 4 (6) | 8 (8) | 5 (5) | 10 (10) | 9 (13) | 11 (14) | 3 (3) | 7 (13)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 3 (3) | 4 (4) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 8 (14) | 7 (10) | 1 (1) | 2 (2) | 2 (3) | 4 (8) | 0 (0) | 7 (9) | 5 (9) | 12 (15) | 13 (16) | 11 (13) | 7 (9) | 31 (39) | 9 (9) | 11 (13)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (11) | 7 (13) | 1 (1) | 2 (4) | 0 (0) | 4 (9) | 1 (1) | 5 (7) | 8 (10) | 10 (13) | 10 (21) | 13 (17) | 9 (10) | 20 (28) | 6 (6) | 11 (18)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 5 (5) | 2 (3) | 2 (2) | 2 (3) | 5 (8)
Duodenogastric Reflux (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 4 (4) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Epigastric Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Gastric Disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Gingival Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hiatus Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperaesthesia Teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired Gastric Emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (4) | 6 (9) | 7 (17) | 3 (7) | 0 (0) | 2 (2) | 4 (6) | 2 (2) | 14 (18) | 10 (12) | 11 (12) | 15 (20) | 13 (19) | 15 (22) | 22 (30) | 6 (7) | 11 (16)
Neutropenic Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Salivary Duct Inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 6 (13) | 7 (11) | 3 (6) | 1 (1) | 0 (0) | 1 (3) | 1 (3) | 6 (6) | 3 (3) | 4 (4) | 6 (10) | 9 (15) | 7 (8) | 15 (21) | 4 (4) | 7 (16)
Application Site Reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Axillary Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 4 (5) | 3 (3) | 1 (1) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 2 (5) | 4 (4) | 2 (2) | 3 (3) | 2 (2) | 5 (5)
Condition Aggravated (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Face Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 2 (3) | 3 (3) | 5 (5) | 8 (10) | 3 (3) | 1 (1) | 1 (2) | 5 (14) | 2 (3) | 15 (15) | 8 (9) | 16 (22) | 14 (22) | 23 (31) | 13 (17) | 31 (37) | 11 (13) | 13 (14)
Feeling Abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait Disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hernia Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza Like Illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Infusion Site Reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Medical Device Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 1 (3) | 3 (3) | 2 (2) | 2 (3) | 4 (6) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Physical Deconditioning (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 5 (6) | 3 (4) | 5 (6) | 0 (0) | 5 (6) | 1 (2) | 7 (7) | 3 (4) | 2 (3)
Soft Tissue Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temperature Intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenderness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination Site Reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Xerosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary Colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic Steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Citrobacter Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis Escherichia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal Oesophagitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes Simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Lung Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Parainfluenzae Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (6)
Pyuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash Pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0)
Tooth Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Urinary Tract Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (5) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 3 (4) | 1 (1) | 3 (3) | 1 (1) | 1 (5) | 1 (1) | 6 (8) | 2 (2) | 1 (1)
Vaginal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post Procedural Discomfort (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post Procedural Swelling (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0
Radiation Necrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon Rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 1 (3) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 6 (6) | 3 (4) | 4 (6) | 6 (9) | 3 (3) | 5 (6) | 10 (11) | 0 (0) | 2 (2)
Amylase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (4) | 3 (6) | 2 (2) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (9) | 3 (4) | 1 (4) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 6 (6) | 2 (2) | 3 (4) | 6 (10) | 3 (3) | 6 (7) | 13 (17) | 0 (0) | 1 (1)
Blood Albumin Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Alkaline Phosphatase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 2 (2)
Blood Bilirubin Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Cholesterol Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Blood Iron Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Lactate Dehydrogenase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Magnesium Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Phosphorus Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Potassium Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Sodium Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Triglycerides Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Urea Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain Natriuretic Peptide Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breath Sounds Abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-reactive Protein Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0)
Electrocardiogram QT Prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 6 (6) | 3 (3) | 0 (0) | 3 (3)
Glomerular Filtration Rate Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International Normalised Ratio Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 3 (4) | 1 (1) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Platelet Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SARS-CoV-2 Test Positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcus Test Positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin T Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin B12 Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 1 (1) | 3 (3) | 3 (3) | 8 (8) | 0 (0) | 13 (13) | 2 (2) | 5 (5)
Weight Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
White Blood Cells Urine Positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 3 (3) | 8 (12) | 2 (5) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 8 (10) | 8 (8) | 5 (6) | 8 (11) | 14 (14) | 7 (7) | 26 (31) | 7 (7) | 12 (16)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Fluid Overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypermagnesaemia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (6) | 2 (4) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Hyperuricaemia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Hypocalcaemia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 4 (4) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 3 (6) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 7 (8) | 2 (2) | 2 (4) | 3 (3) | 3 (5) | 2 (2) | 12 (17) | 3 (5) | 3 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 2 (2) | 0 | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 3 (4) | 0 (0) | 3 (3) | 2 (2) | 10 (20) | 1 (2) | 3 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (4) | 1 (1) | 2 (2) | 2 (2) | 6 (11) | 2 (3) | 4 (6)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 4 (7) | 2 (2) | 0 (0)
Iron Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (6) | 1 (1) | 3 (3) | 7 (9) | 6 (6) | 2 (3) | 8 (13) | 2 (2) | 5 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (6) | 0 (0) | 4 (4) | 1 (1) | 6 (6) | 2 (2) | 9 (10) | 1 (1) | 3 (4)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Muscle Tightness (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 4 (6) | 4 (5) | 5 (6) | 4 (4) | 3 (3) | 4 (4) | 5 (6) | 3 (3)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 5 (6) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 2 (2)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Amputation Stump Pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Autonomic Nervous System Imbalance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autonomic Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Balance Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carpal Tunnel Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed Level of Consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disturbance in Attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 5 (5) | 3 (3) | 4 (5)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (5) | 6 (7) | 0 (0) | 2 (2) | 0 (0) | 5 (5)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 4 (5) | 5 (11) | 5 (6) | 5 (7) | 4 (4) | 4 (10)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Metabolic Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mononeuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Monoplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 5 (6) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Neurotoxicity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Paresis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral Motor Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Peripheral Sensorimotor Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (6) | 2 (4) | 1 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 9 (14) | 2 (3) | 4 (4) | 7 (11) | 11 (14) | 6 (6) | 11 (11) | 3 (3) | 7 (7)
Peroneal Nerve Palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyramidal Tract Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless Legs Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal Cord Compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Taste Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed Mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucination, Olfactory (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination, Visual (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 5 (5) | 5 (5) | 8 (8) | 3 (3) | 7 (7)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bladder Discomfort (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Calculus Bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertonic Bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urge Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perineal Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal Discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal Dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0
Vulvovaginal Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adductor Vocal Cord Weakness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 3 (3) | 5 (6) | 2 (2) | 5 (5) | 2 (3) | 3 (10)
Dysaesthesia Pharynx (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 4 (4) | 2 (3) | 6 (8) | 6 (7) | 10 (12)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (3)
Paranasal Sinus Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper-airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasomotor Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 5 (5) | 7 (7) | 8 (9) | 3 (3) | 9 (9) | 14 (14) | 2 (2) | 6 (6)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis Bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hair Texture Abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lichenoid Keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail Discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail Dystrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 2 (2)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 4 (4) | 1 (2) | 6 (7) | 3 (4) | 6 (7) | 1 (1) | 3 (3)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 5 (5) | 2 (2) | 6 (7) | 3 (4) | 3 (5)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash Macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot Flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 4 (4) | 1 (1) | 3 (9) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 7 (7) | 0 (0) | 1 (1)
Jugular Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis Superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular Compression (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
No participants with castration-resistant prostate cancer were enrolled, hence no prostate-specific antigen (PSA) data were available and pre-specified outcome measure related to PSA data are not reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is at least 12 months but less than 18 months from the end of study (database lock). The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT02988817/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT02988817/SAP_001.pdf